CLINICAL TRIAL: NCT02583152
Title: Use of New Imaging Technology to Assess Effect of Enzyme Replacment Therapy on Eye Disease Progession in Mucopolysacchardiosis
Brief Title: New Imaging Technology to Assess Effect of Enzyme Replacment Therapy on Eye Disease Progession in Mucopolysacchardiosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manchester Royal Eye Hospital (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: R04002
Record Dates: First submitted 2015-09-10; First posted 2015-10-22 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Mucopolysaccharidoses
MeSH Terms: conditions — Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MPS patient cohort: Participants with Mucopolysaccharidosis. types I-IV, VI and VII will be recruited from the paediatric and adult ophthalmology. Participants over the age of three who are able to comply and be investigated.

SUMMARY:
Mucopolysaccharidoses (MPS) are currently treated with Enzyme replacement therapy and Bone Marrow Transplantation (BMT). No current evidence on the effectiveness on these therapies on the eye in this systemic disease is avalible. Using new imaging techniques; previously subjective data can be quantified and compared to determine if there is an improvment in the vision of patients with MPS.

DETAILED DESCRIPTION:
The mucopolysaccharidoses (MPS) are a group of hereditary disorders which arise from defects in enzymes which break down glycosaminoglycans (GAGs) which occur in a wide variety of tissues, resulting in multiple systemic complications. Sight loss occurs in MPS due to corneal clouding, retinal degeneration, glaucoma and damage to the optic nerve. Corneal opacification occurs in infancy in several MPS subtypes and in the untreated disease the opacification is thought to be progressive, contributing to significant visual impairment in many patients. Improvements in quality of life and lifespan as a result of early treatment (with enzyme replacement therapy and haematopoetic stem cell transplantation) have meant that management of ocular complications and preservation of vision has increased importance.

A repeatable, reliable technique for quantification of corneal clouding will allow objective demonstration of the effect of treatments such as ERT in stabilisation or improvement of corneal clouding, and to establish the natural history of corneal opacification in MPS.

The investigators have previously developed the Iris camera (Irisguard Corp, McLean, VA 22102, USA) technology to give an objective measure of corneal clouding (Irisguard model IGAD100 ®) (Aslam et al 2009). The investigators demonstrated that use of the iris camera for corneal opacification assessment in MPS is feasibile, practical and has shown evidence for validity and reliability (Aslam et al 2012) (research funded in part by Biomarin Europe Ltd). The densitometry program for the Pentacam® Scheimpflug camera has also been shown to be able to provide measurements of corneal clouding in MPS .This research proposal will allow us to use to these techniques to quantify corneal clouding over time in MPS patients and to assess the effects of treatment with ERT and HSCT on corneal opacification.

ELIGIBILITY:
Inclusion Criteria:

* Adult and paediatric participants with MPS and corneal opacification will be potentially eligible for this study, including those untreated, treated with previous haematopetic stem cell transplant, and treated with ERT.
* Participants who have a confirmed diagnosis of mucopolysaccharosisis type I (Hurler, Hurler/Scheie and Scheie), MPS type II (Hunter), type III (Sanfilippo) type IV (Morquio) and type VI (MaroteauxLamy), type VII (Sly) will be potentially eligible. In order to cooperate with the examinations, the participant needs to be able to hold relatively still while seated at an instrument with a head rest and hold fixation for several seconds for this reason participants over the age of 3 years will be eligible.

Exclusion Criteria:

* Those who are aged under 3 years or who have significant neurological involvement which would influence understanding and/or cooperation.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Adult and paediatric participants with MPS and corneal opacification will be potentially eligible for this study, including those untreated, treated with previous haematopetic stem cell transplant, and treated with ERT.
  * Participants who have a confirmed diagnosis of mucopolysaccharosisis type I (Hurler, Hurler/Scheie and Scheie), MPS type II (Hunter), type III (Sanfilippo) type IV (Morquio) and type VI (MaroteauxLamy), type VII (Sly) will be eligible if able to hold relatively still while seated at an instrument with a head rest.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Corneal densitometry scores in participants on treatment | 60 months study period

SECONDARY OUTCOMES:
Corneal clouding score over time in patients on treatment. | 60 months study period

OTHER OUTCOMES:
Repeatability and accessibility for each imaging technique | 60 months study period
Retinal morphology changes with Optos wide field digital imaging and high resolution OCT | 60 months study period

CONTACTS AND LOCATIONS:
Overall Officials: Jane Ashworth, MBChB, PhD, Principal Investigator — Central Manchester Foundation Trust
Locations (1):
- Manchester Royal Eye Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No